CLINICAL TRIAL: NCT04078932
Title: Getting Real About The Talk (GReAT) Project
Brief Title: The Getting Real About The Talk (GReAT) Project - A Qualitative, Patient-Centered Evaluation of the Factors for Successfully Having 'The Talk' and Implementation for Attending and Trainee Physicians
Acronym: GReAT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jeffrey Eugene, MD (Other)
Collaborators: Accreditation Council for Graduate Medical Education (Other)
Responsible Party: Sponsor-Investigator, Jeffrey Eugene, MD, Physician, Adolescent Medicine Fellow, Post Graduate Year (PGY)-6, University of Pennsylvania
Organization: University of Pennsylvania (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: GDNJJESC139
Record Dates: First submitted 2019-08-28; First posted 2019-09-06 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Self Efficacy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Cohort of residents trained in the conversation script who will utilize the script at pediatric clinic visits. Will evaluate baseline feelings of comfort and self-efficacy prior to being trained in the script (pre-intervention measures). After being trained in the conversation script (the intervention), the following will be measured (post-intervention measures): frequency of facilitating conversations on safely navigating police encounters in clinical practice, feelings of comfort and self-efficacy.
  Interventions: Behavioral: Violence Prevention Conversation Script to Discuss Safely Navigating Police Encounters
- Control (No Intervention): Cohort of residents at another clinical site with a similar community demographic make-up who do not receive the intervention. In the control group, we will measure frequency of facilitating conversations on safely navigating police encounters in clinical practice, feelings of comfort and self-efficacy.

INTERVENTIONS:
Behavioral: Violence Prevention Conversation Script to Discuss Safely Navigating Police Encounters — A conversation script to facilitate conversations on safely navigating police encounters as anticipatory guidance and violence prevention strategy. The conversation script will be created using expert recommendations from existing resources and using recommendations (determined from focus groups) from black male youth and their caregivers. The script will be patient-centered.
  Arms: Intervention

SUMMARY:
The killing of young black men by police officers is a major public health issue and is a clear health disparity. Black men are 21 times more likely to be fatally shot by a police officer than white men. Homicide is the second-leading cause of death of black males, ages 15-34. It is disconcerting to consider that this statistic includes homicide by police officer. Pediatricians have an opportunity to contribute to violence prevention efforts and social justice advocacy for young black men in regards to interactions with police officers.

We seek to engage residents in social justice advocacy by preparing them to discuss safely navigating police encounters with young black males. Adverse police encounters can result in poor mental health outcomes, physical trauma, and death. We will develop a conversation script with input from existing expert resources, black male youth, and their caregivers. The script will be patient-centered and will be used to facilitate a conversation about safely navigating encounters with police officers. Utilizing a train-the-trainer model, attending pediatric physicians will be trained to use the script in their practice as well as model and demonstrate how to use the script for pediatric residents. We hypothesize that pediatric residents trained in the conversation script will be empowered to facilitate discussions on safely navigating police encounters in the primary care clinic setting and will exhibit increased comfort and greater levels of self-efficacy from baseline measures.

ELIGIBILITY:
Inclusion Criteria:

* Resident physician trainee at a designated academic medical center-based primary care clinic serving predominately black youth in Philadelphia

Exclusion Criteria:

* Non-resident physician trainee
* Resident physician preference to not participate
* Not affiliated with the designated academic medical center-based primary care clinic

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-12-01 (Estimated); Primary Completion 2022-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Resident physician Self-Efficacy | Change from Baseline Feelings of Self-Efficacy at 6 months
  Likert-type, self-reported Self-efficacy instrument. The items on the survey instrument will assess for feelings of self-efficacy pre-intervention (baseline) and 6 months post-intervention. Respondents will select their level of agreement with each item on the survey, selecting within a range from "strongly disagree" to "strongly agree". "Strongly agree" indicates the highest level of agreement with each statement on the survey. Respondents who predominately select "strongly agree" for the items on the survey express greater levels of self-efficacy with delivering the intervention.

SECONDARY OUTCOMES:
Resident physician Comfort Level | Change from Baseline Comfort Level at 6 months
  Likert-type, self-reported instrument assessing comfort with delivering the intervention. The items on the survey instrument will assess for comfort pre-intervention (baseline) and 6 months post-intervention. Respondents will select their level of agreement with each item on the survey, selecting within a range from "strongly disagree" to "strongly agree". "Strongly agree" indicates the highest level of agreement with each statement on the survey. Respondents who predominately select "strongly agree" for the items on the survey express greater levels of comfort with delivering the intervention.
Frequency of delivering the script in clinical practice | Change from Baseline Frequency of Delivering the Script at 6 months
  Self-response to the following question: In the past 6 months, how many times have you delivered the conversation script (the intervention) to African-American male youth ages 9-18? Respondents will answer by selecting between the following choices: 0 times, 1-5 times, 5-10 times, 10-15 times, and greater than 15 times.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] 1.ACLU. "Know your rights: what to do if you're stopped by police, immigration agents or the FBI". https://www.aclu.org/know-your-rights/what-do-if-youre-stopped-police-immigration-agents-or-fbi. Updated 2019. Accessed February 23, 2019.
- [Background] Allen, VD and Solomon, P. 'EVIP-Edutainment Violence Intervention/Prevention Model'. Journal of Human Behavior in the Social Environment, 2016. 26.(3,4). 325-335
- [Background] Boyd RW, Ellison AM, Horn IB. Police, Equity, and Child Health. Pediatrics. 2016;137(3):e20152711. Pediatrics. 2018 Jul;142(1):e20181137. doi: 10.1542/peds.2018-1137. No abstract available. PMID 29959175
- [Background] Boynton-Jarrett R, Ryan LM, Berkman LF, Wright RJ. Cumulative violence exposure and self-rated health: longitudinal study of adolescents in the United States. Pediatrics. 2008 Nov;122(5):961-70. doi: 10.1542/peds.2007-3063. PMID 18977974
- [Background] Bui AL, Coates MM, Matthay EC. Years of life lost due to encounters with law enforcement in the USA, 2015-2016. J Epidemiol Community Health. 2018 Aug;72(8):715-718. doi: 10.1136/jech-2017-210059. Epub 2018 May 7. PMID 29735570
- [Background] Centers for Disease Control and Prevention (CDC). Leading Causes of Death (LCOD) by Age Group, Black Males-United States, 2015. Office of Minority Health and Health Equity. https://www.cdc.gov/healthequity/lcod/men/2015/black/index.htm. 2019. Accessed May 3, 2019.
- [Background] Charles D, Himmelstein K, Keenan W, Barcelo N; White Coats for Black Lives National Working Group. White Coats for Black Lives: Medical Students Responding to Racism and Police Brutality. J Urban Health. 2015 Dec;92(6):1007-10. doi: 10.1007/s11524-015-9993-9. No abstract available. PMID 26382654
- [Background] Dare to Be King. "Navigating encounters with police." http://daretobeking.net/tta/nep/. 2019. Accessed February 23, 2019.
- [Background] Gabrielson R, Grochowski Jones R, Sagara E. Deadly force, in black and white. 2014. Available at: https:// www.propublica. org/ article/ deadly- force- in black-and- white. Accessed February 23, 2019
- [Background] Geller A, Fagan J, Tyler T, Link BG. Aggressive policing and the mental health of young urban men. Am J Public Health. 2014 Dec;104(12):2321-7. doi: 10.2105/AJPH.2014.302046. Epub 2014 Oct 16. PMID 25322310
- [Background] 11.Get Home Safely: 10 Rules of Survival. http://www.pbs.org/black-culture/connect/talk-back/10_rules_of_survival_if_stopped_by_police/. Accessed on February 23, 2019
- [Background] Maroney T, Zuckerman B. "The Talk," Physician Version: Special Considerations for African American, Male Adolescents. Pediatrics. 2018 Feb;141(2):e20171462. doi: 10.1542/peds.2017-1462. Epub 2018 Jan 9. No abstract available. PMID 29317517
- [Background] Raja Staggers-Hakim. The nations unprotected children and the ghost of Mike Brown, or the impact of national police killings on the health and social development of African American boys. Journal of Human Behavior in the Social Environment.
- [Background] Sege RD, Hatmaker-Flanigan E, De Vos E, Levin-Goodman R, Spivak H. Anticipatory guidance and violence prevention: results from family and pediatrician focus groups. Pediatrics. 2006 Feb;117(2):455-63. doi: 10.1542/peds.2005-0377. PMID 16452366
- [Background] Young black men killed by US police at highest rate in year of 1,134 deaths. The Guardian. https://www.theguardian.com/us-news/2015/dec/31/the-counted-police-killings-2015-young-black-men. Published online 31 Dec 2015. Accessed on February 24, 2019
- [Background] Bandura, Albert. Guide for Constructing Self-Efficacy Scales (book chapter). Self-Efficacy Beliefs of Adolescents, edited by Frank Pajares and Tim Urdan, Information Age Publishing (IAP), Inc. 2006.
- [Background] Mapping Police Violence. https://mappingpoliceviolence.org. Updated January 2, 2019. Accessed on February 25, 2019
- [Background] Sherer M, et al. The Self-Efficacy Scale: Construction and Validation. Psychological Reports, 1982, 51, 663-671.